CLINICAL TRIAL: NCT02526173
Title: A Prospective Randomized Clinical Trial Using Dehydrated Human Amnion/Chorion Membrane (dHACM) in Nerve Sparing Robotic Assisted Laparoscopic Radical Prostatectomy (RALP) - Effect on Potency Outcomes
Brief Title: DHACM in Robotic Assisted Laparoscopic Prostatectomy (RALP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFRLP003
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- dHACM (Experimental): This group will receive RALP using full nerve sparing technique plus dHACM application.
  Interventions: Procedure: RALP using full nerve sparing technique; Other: dHACM Application
- Control (Other): This group will receive RALP using full nerve sparing technique only.
  Interventions: Procedure: RALP using full nerve sparing technique

INTERVENTIONS:
Procedure: RALP using full nerve sparing technique — RALP using full nerve sparing technique
Other: dHACM Application — 2x12 sheet of dHACM applied to the neurovascular bundle
  Other Names: HCT/P Part 361
  Arms: dHACM

SUMMARY:
The investigators will examine the beneficial impacts of applying of dHACM on the preserved neurovascular bundles (cavernosal nerves) and the prostate bed during robotic assisted laparoscopic prostatectomy. Such application can result in promotion of soft tissue healing and reduction of inflammation at the operative site and thus an acceleration of return of potency regulating cavernosal nerves.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the effectiveness of dehydrated human amnion/chorion membrane (dHACM) in reducing neurovascular bundle inflammation in prostate cancer patients undergoing bilateral full nerve sparing robotic assisted laparoscopic radical prostatectomy (RALP). Specifically, this study compares potency outcomes in patients who had full nerve sparing RALP procedures with dHACM application to the neurovascular bundles to that of full nerve sparing RALP without dHACM application to neurovascular bundles.

Patients will be randomized to one of two possible treatment groups:

* Group 1 - Treatment Group ( Full Nerve Sparing RALP + AmnioFix®)
* Group 2 - Control Group ( Full Nerve Sparing RALP alone)

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between the ages 40-70.
2. Primary diagnosis of prostate cancer requiring surgical intervention
3. Have a willingness to comply with follow-up examination
4. Have ability to provide full written consent
5. Primary diagnosis of untreated with clinically localized prostate cancer with Gleason score of 6, 7,8 or 9
6. Planned elective radical prostatectomy with bilateral full nerve sparing technique
7. Patients who currently have a pre-operative SHIM > 19
8. Negative urinalysis within 7 days prior to date of surgery

Exclusion Criteria:

1. Has signs or symptoms of any other disease which could result in allograft failure, or has experienced graft failure in the past
2. Has any condition(s), which seriously compromises the subject's ability to participate in this study, or has a known history of poor adherence with medical treatment
3. Has comorbid conditions that can be confused with or can exacerbate the condition, including diabetes or Advanced atherosclerotic vascular disease
4. Is unable to sign or understand informed consent
5. Is unable to comply with penile rehabilitation, including oral 5-phosphodiesterase inhibitor
6. Has a history of drug or alcohol abuse within last 12 months
7. Has autoimmune disease or a known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV
8. Is allergic to Aminoglycoside antibiotics (such as Gentamicin and/or Streptomycin)
9. Patients with a history of more than two weeks treatment with immuno-suppressants (including systemic corticosteroids), cytotoxic chemotherapy within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study
10. Patients currently enrolled in another study. Concurrent enrollment in another study is prohibited
11. Has had prior hormonal therapy such as Lupron or oral anti-androgens
12. Living outside of United States
13. Partial nerve sparing technique used during Radical Prostatectomy

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Potency as assessed by Sexual Health Inventory for Men (SHIM) Score | 12 months
  As measured by SHIM
Return to sexual function | 12 months
  Patient directed questionnaire

SECONDARY OUTCOMES:
Continence | 12 months
  As assessed by American Urological Association (AUA) score
Continence | 12 months
  Patient directed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vipul Patel, MD, Principal Investigator — MiMedx Group, Inc.
Locations (1):
- Florida Hospital: Global Robotics Institute, Celebration, Florida, United States